CLINICAL TRIAL: NCT00831116
Title: Chemometric Observation of Lipid Core Plaques of Interest in Native Coronary Arteries Registry
Brief Title: An Observational Study of Cholesterol in Coronary Arteries
Acronym: COLOR
Status: Completed | Type: Observational
Sponsor: Infraredx (Industry)
Responsible Party: Sponsor
Other Study IDs: 0111
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Myocardial Infarction; Angina; Coronary Artery Disease; Myocardial Ischemia
Keywords: near infrared spectroscopy; LipiScan; lipid core; percutaneous coronary intervention; myocardial infarction; NIRS; intravascular imaging
MeSH Terms: conditions — Myocardial Infarction; Angina Pectoris; Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- LipiScan: Subjects who have at least one native coronary artery imaged with the LipiScan CIS.
  Interventions: Device: Intravascular Near Infrared Spectroscopy

INTERVENTIONS:
Device: Intravascular Near Infrared Spectroscopy — Intravascular imaging with a catheter based spectroscopy system.
  Other Names: LipiScan Coronary Imaging System

SUMMARY:
In April 2008, a coronary catheter based imaging system, LipiScan, was cleared by the FDA for use in detecting lipid core containing containing plaques of interest (LCP). These plaques are rich in cholesterol. The way that cholesterol and other lipids deposit with the coronary artery is unique to each patient. This study is an organized attempt to observe the LCP and the variety of ways that it presents in patients as detected by this recently approved device. This information will be used for physician training and to observe the behavior of the LCP in response to no therapy and currently approved therapies. The purpose of this project is further medical knowledge of the LCP and its treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age.
* Subject is scheduled for elective coronary catheterization.
* LipiScan CIS, LipiScan IVUS Imaging System, or TVC Imaging System use is not contra-indicated.
* At least one chemogram from a native coronary artery is available for submission to the registry.
* Able to read, understand and sign the informed consent.

Exclusion Criteria:

* Subject is pregnant or nursing.
* Subject life expectancy is less than 2 years at time of index catheterization.
* All submitted chemograms are obtained with the LipiScan, LipiScan IVUS, or TVC(R) Imaging Catheter positioned within a coronary artery bypass graft.
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from those presenting or referred to the cardiac catheterization laboratory for elective cardiac catheterization.
Sampling Method: Non-Probability Sample
Enrollment: 2067 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Identify associations of LCP with angiographic or symptomatic presentation of coronary artery disease in a catheterization laboratory population | after completion of the study - during data analysis

SECONDARY OUTCOMES:
Identification of associations that LCP or the Lipid Core Burden Index (LCBI) may have with atherosclerosis appearance, progression, regression, and/or cardiac event | Upto 2 years post procedure(baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Giora Weisz, MD, Study Chair — Columbia University
Locations (22):
- United States (22):
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - Scottsdale Healthcare, Scottsdale, Arizona
  - University of California, Los Angeles Medical Center, Los Angeles, California
  - University of California Irvine Medical Center, Orange, California
  - San Francisco Veterans Affairs Medical Center, San Francisco, California
  - University of Florida, Gainesville, Gainesville, Florida
  - Pepin Heart Hospital, Tampa, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - Crittenton Shelton Heart Center:, Rochester Hills, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Saint Louis University Hospital, St Louis, Missouri
  - Mount Sinai School of Medicine, New York, New York
  - Columbia Universtiy Medical Center, New York, New York
  - Pinnacle Heart & Vascular Institute, Harrisburg, Pennsylvania
  - Medical University of South Carolina Hospital, Charleston, South Carolina
  - Veterans Affairs, North Texas Health Care Systems, Dallas, Texas
  - Swedish Medical Center, Seattle, Washington